CLINICAL TRIAL: NCT01258673
Title: A Randomized, Double-blind, Multicenter Clinical Study to Evaluate Efficacy and Safety of Fimasartan/Hydrochlorothiazide Combination-therapy in Comparison With Fimasartan Monotherapy for Essential Hypertension Patients Not Controlled by Fimasartan 60mg(Phase 3)
Brief Title: A Clinical Study to Evaluate Efficacy and Safety of Fimasartan/Hydrochlorothiazide Combination-therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Seoul National University Hospital (Other); The Catholic University of Korea (Other); Korea University Guro Hospital (Other); DongGuk University (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other); Gangnam Severance Hospital (Other); Severance Hospital (Other); Ajou University (Other); Chonbuk National University Hospital (Other); Cheil General Hospital and Women's Healthcare Center (Other); Chonnam National University Hospital (Other); Hanyang University Guri Hospital (Other); Yonsei University (Other); Ilsan-Paik Hospital (Unknown); SMG-SNU Boramae Medical Center (Other); Kyung Hee University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-FHC-CT-301
Record Dates: First submitted 2010-12-10; First posted 2010-12-13 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2010-12

CONDITIONS: Essential Hypertension
Keywords: Fimasartan; Fimasartan/Hydrochlorothiazide combination
MeSH Terms: conditions — Essential Hypertension | interventions — fimasartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fimasartan/HCTZ combination group (Experimental)
  Interventions: Drug: Fimasartan/HCTZ combination
- Fimasartan group (Active Comparator)
  Interventions: Drug: Fimasartan

INTERVENTIONS:
Drug: Fimasartan/HCTZ combination — Fimasartan/HCTZ combination 60/12.5mg 120/12.5mg
  Arms: Fimasartan/HCTZ combination group
Drug: Fimasartan — Fimasartan 60mg, 120mg
  Arms: Fimasartan group

SUMMARY:
The purpose of this study is to evaluate the antihypertensive efficacy and safety of Fimasartan/Hydrochlorothiazide combination 60/12.5mg~120/12.5mg in patients with essential hypertension who are not controlled by fimasartan 60mg.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 years of age and older
* Patients with antihypertensive agents at screening: DBP<110mmHg or Patients without antihypertensive agents at screening: DBP 90mmHg~120mmHg
* Subjects who agree to participate in this sudy and give written informed consent
* Subjects considered to understand the study, be cooperative, and able to be followed-up until the end of the study
* Patients with not controlled blood pressure at baseline visit, by fimasartan 60mg 4weeks treatment, DBP 90mmHg~109mmHg and SBP<180mmHg

Exclusion Criteria:

* The sitting DBP is more than 120mmHg or severe hypertensive patient with sitting systolic blood pressure over 200mmHg Patients with secondary hypertension
* Patients who are measured the mean difference of mean blood pressure under SiDBP 10mmHg or SiSBP 20mmHg at screening or baseline visit
* Patients with severe renal(Creatinine more 1.5 times than upper limit of normal), gastrointestinal, hematological or hepatic(AST, ALT more 2 twice more than upper limit of normal)disease etc. which might affect absorption, disposition, metabolism or excretion of the drug
* Patients with postural hypotension
* Patients with sever insulin dependent diabetes mellitus or uncontrolled diabetes mellitus(HbA1c>9%, regimen change of oral hypoglycemic agents within 12weeks, treated insulin before screening)
* Patients with a history of myocardial infarction, severe coronary artery disease or clinically significant heart failure or valvular defect in last 6 months
* Patients with consumptive disease, autoimmune disease, connective tissue disease
* Patients with a history of type B or C hepatitis(include carrier)
* Patients with HIV or hepatitis
* Patients with clinically significant laboratory abnormality
* Patients receiving any drugs known to affect blood pressure or medical treatments that can influence the blood pressure
* Patients with allergy or contraindication to any angiotensin II receptor antagonists
* Female of childbearing potential who does not undergo hysterectomy or is not post-menopausal
* Patients judged to have a history of alcohol or drug abuse by the investigator
* Patients participated other clinical trial 12 weeks before Screening - Patients judged to be inappropriate for this study by the investigator with other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Diastolic Blood Pressure | 4week

SECONDARY OUTCOMES:
Systolic Blood Pressure / Diastolic Blood Pressure | 4week, 8week / 8week

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Bundang, Sungnam, South Korea

REFERENCES:
- [Derived] Rhee MY, Baek SH, Kim W, Park CG, Park SW, Oh BH, Kim SH, Kim JJ, Shin JH, Yoo BS, Rim SJ, Ha JW, Doh JH, Ahn Y, Chae JK, Park JB, Kim SK, Kim CH. Efficacy of fimasartan/hydrochlorothiazide combination in hypertensive patients inadequately controlled by fimasartan monotherapy. Drug Des Devel Ther. 2015 Jun 2;9:2847-54. doi: 10.2147/DDDT.S82098. eCollection 2015. PMID 26082615
- [Derived] Fimasartan. Am J Cardiovasc Drugs. 2011 Aug 1;11(4):249-52. doi: 10.2165/11533640-000000000-00000. PMID 21740078